CLINICAL TRIAL: NCT01682655
Title: The Influence of Apolipoprotein C3 Variants on Liver Steatosis and Serum Liver Enzyme Values in Obese Children
Brief Title: Genetic Variant in Apolipoprotein C3 Gene and Fatty Liver in Obese Children
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 101015-F
Record Dates: First submitted 2012-09-03; First posted 2012-09-11 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2013-11

CONDITIONS: Fatty Liver; Obesity
MeSH Terms: conditions — Fatty Liver; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, WBC DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In the past decades, obesity in children is much more prevalent in the world. Given the increasing prevalence of pediatric obesity worldwide, fatty liver incidence is on the rise.

Genetic variant in apolipoprotein C3 (APOC3) gene is associated with increased liver fat content in adults.

The aim of this study is to find out whether APOC3 single nucleotide polymorphism (SNP) influence fatty liver in obese children and adolescent.

DETAILED DESCRIPTION:
The primary aim of this study is to assess the associations between to investigate the association of rs2854117 C > T and rs2854116 T > C SNPs of the APOC3 gene with liver steatosis, as measured by liver ultrasound.

As a secondary aim, the investigators will examine the associations between APOC3 rs2854117 C > T and rs2854116 T > C SNPs and serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels. In addition, the investigators will further analyze the association with other biomarkers, such as body mass index, adiponectin and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-18 years old
* Obesity definition: BMI > 95% according to the age- and gender-specific standard suggested by National Health Institute in Taiwan
* Willing to give written informed consent by parents

Exclusion Criteria:

* Alcohol consumption
* Chronic liver diseases, including hepatitis B, hepatitis C, Wilson disease and autoimmune hepatitis
* Major systemic diseases, including cardiopulmonary disease, renal failure, cancer, and psychotic disorder

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Obese children and adolescents in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
genotype distribution of APOC3 rs2854117 and rs2854116 polymorphisms in subjects with and without liver steatosis | Oct 2013 ~ Dec 2014

SECONDARY OUTCOMES:
genotype distribution of APOC3 rs2854117 and rs2854116 polymorphisms in subjects with and without insulin resistance | Oct 2013 ~ Dec 2014

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Cheng Lin, MD, PhD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan, Taiwan